CLINICAL TRIAL: NCT01215617
Title: The Effect of Aerobic Interval Training on Obstructive Sleep Apnea, Cardiovascular and Pulmonary Function in Obese Patients
Brief Title: The Effect of Aerobic Interval Training on Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2010/1539-5; 20101539-2 (Other: REK)
Record Dates: First submitted 2010-10-04; First posted 2010-10-06 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Randomized controlled study; Exercise training; Lung function; Heart function
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Interval Training (Experimental): Patients randomized to training will meet for supervised aerobic interval training three times per week for 3 months. The interval training session consists of 10 minutes warm up and continues with 4 x 4 minutes of high intensity intervals at 90-95% of maximal heart rate
  Interventions: Behavioral: Aerobic Interval training
- Control (Other): Patients will receive standard medical treatment at the University Hospital lung department.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Aerobic Interval training — Treadmill walking or running - 3 times per week for 3 months. The interval training session consists of 10 minutes warm up and continues with 4 x 4 minutes high intensity intervals at 90-95% of maximal heart rate. Training intensity will be supervised through the use of Polar pulse monitors and the BORG scale of subjective perceived exhaustion.
  Arms: Aerobic Interval Training
Behavioral: Control — Standard medical treatment
  Arms: Control

SUMMARY:
The purpose of this study is to investigate if 3 months of interval training improves obstructive sleep apnea in obese patients diagnosed with moderate to severe obstructive sleep apnea. The working hypothesis is that 3 months of 3 weekly aerobic interval training sessions improve obstructive sleep apnea and sleep quality in obese patients.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) is characterized by repetitive obstruction and collapse of the upper airway resulting in successive episodes of cessation of or decreased respiratory airflow, causing oxygen desaturation, awakening, loud snoring and daytime sleepiness in patients. Sleep apnea is frequently associated with co-morbidity such as obesity, diabetes, hypertension, the metabolic syndrome and cardiovascular disease. Lack of exercise is associated with OSAS severity, independent of body mass. Participation and motivation to exercise is low in OSAS patients, with less that one third of the patients reporting regular exercise routines. We aim to investigate if aerobic interval training improves OSAS in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30 kg/M2
* Apne - hypopnea index (AHI) > 10
* No significant comorbidities
* Abel to exercise

Exclusion Criteria:

* Inability to exercise due to musculoskeletal conditions
* Known ischemic cardiovascular disease
* Drug abuse
* Mental illnesses

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index change | Baseline, 3 and 6 months
  Measured by Polysomnography

SECONDARY OUTCOMES:
Sleep quality | Baseline, 3 and 6 months
  Epworth Sleepiness Scale

CONTACTS AND LOCATIONS:
Overall Officials: Trine Karlsen, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Karlsen T, Nes BM, Tjonna AE, Engstrom M, Stoylen A, Steinshamn S. High-intensity interval training improves obstructive sleep apnoea. BMJ Open Sport Exerc Med. 2017 Feb 8;2(1):bmjsem-2016-000155. doi: 10.1136/bmjsem-2016-000155. eCollection 2016. PMID 29616142